CLINICAL TRIAL: NCT05315323
Title: Clinical Use of EVUSHELD as Pre-exposure Prophylaxis in Real-world Setting - A Multi-center Observational Prospective Study to Determine Utilization and Clinical Outcomes of EVUSHELD in Gulf Cooperation Council Countries
Brief Title: Clinical Use of EVUSHELD as Pre-exposure Prophylaxis in Real-world Setting in Gulf Cooperation Council Countries
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8851R00001
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; AZD7442; EVUSHELD; Real-world Setting
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study on Clinical Use of EVUSHELD (AZD7442) as Pre-exposure Prophylaxis in the Real-world Setting - A Multi-Centre Observational Prospective Study to Determine the Utilization and Clinical Outcomes of EVUSHELD in Gulf Cooperation Council Countries

DETAILED DESCRIPTION:
Study on Clinical use of EVUSHELD (AZD7442) as pre-exposure prophylaxis in the Real-world Setting Observational Prospective Study to determine the utilization and Clinical Outcomes of EVUSHELD in GCC.

This will be a multi-country, multi-centre, single-arm, observational, prospective study using primary data collection to describe the demographic and clinical characteristics of patients who received the first dose of AZD7442 for the prevention of SARS-CoV-2 infection causing symptomatic COVID-19 illness. The study will be conducted in the hospital/centers that are authorized to administer AZD7442, agree to participate in the study, and wherein investigators have access to all medical records (electronic/paper) for individual patients. The physicians at the hospital/centers will make a decision to administer AZD7442 to patients according to the local regulations (including the prescribing information) and such a decision to use AZD7442 is independent of the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving their first dose of AZD7442 for the prevention of SARS-CoV-2 infection within the 30 days prior to study enrolment.
* The ability or willingness to sign informed consent/assent forms

Exclusion Criteria:

* Patients currently participating in interventional clinical trials of SARS-CoV-2 vaccines, other SARS-CoV-2 prophylactic interventions, or COVID-19 treatments.
* Patients with an ongoing COVID-19 infection at the time of AZD7442 administration as judged by the study physician.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants included in this this study are all individuals who have received a AZD7442 first ever dose for the prevention of SARS-CoV-2 infection. In most countries this will be primarily subjects aged 12+ years.
Sampling Method: Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Demographics | 12 month
  To describe the baseline demographic of individuals receiving AZD7442 for pre-exposure prophylaxis
clinical characteristics | 12 month
  To describe the clinical characteristics of individuals receiving AZD7442 for pre-exposure prophylaxis
baseline and repeat administration | 12 month
  To describe the baseline and repeat administration(s) of AZD7442 for prevention of SARS-CoV-2 infection

SECONDARY OUTCOMES:
Incidence of SARS-CoV-2 infection | 12 Month
  To describe the incidence of SARS-CoV-2 infection (asymptomatic or symptomatic), medically attended COVID-19, and COVID-19 related hospitalization and death up to 12 months after administration of AZD7442 for prevention of SARS-CoV-2 infection
Incidence of all-cause hospitalization and mortality | 12 Month
  To describe the incidence of all-cause hospitalization and mortality during the 12 months after administration of AZD7442 for prevention of SAR-CoV-2 infection
COVID-19 risk behavior at time of AZD7442 | 12 Month
  To describe COVID-19 risk behavior at the time of AZD7442 injection and during the 12 months after first administration of AZD7442 for prevention of SARS-CoV-2 infection
Describe health-related quality of life | 12 Month
  To describe health-related quality of life (QoL) at the time of AZD7442 first injection and during the 12 months after first administration of AZD7442 for prevention of SARS-CoV-2 infection
describe COVID-19-related healthcare resource utilization | 12 Month
  To describe COVID-19-related healthcare resource utilization during the 12 months after first administration of AZD7442 for prevention of SARS-CoV-2 infection

OTHER OUTCOMES:
Describe the demographic and clinical characteristics | 12 Month
  To describe the demographic and clinical characteristics of SARS-CoV-2 infection (asymptomatic or symptomatic), medically attended COVID-19, and COVID-19 related hospitalized cases occurring up to 12 months following AZD7442 first administration for prevention of SARS-CoV-2 infection in comparison to non-cases
Describe the incidence of long COVID syndrome | 12 Month
  To describe the incidence of long COVID syndrome following AZD7442 administration for prevention of SARS-CoV-2 infection
Describe all-cause HCRU | 12 Month
  To describe all-cause HCRU in the 12 months prior to and during the 12 months after AZD7442 first injection for prevention of SARS-CoV-2 infection
Describe COVID-19-related work loss/school absenteeism | 12 Month
  To describe COVID-19-related work loss/school absenteeism at baseline (last 6 months) and during the 12 months after first administration of AZD7442 for prevention of SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Locations (2):
- United Arab Emirates (2):
  - Research Site, Abu Dhabi
  - Research Site, Dubai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ is accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
  For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Url Preview for AstraZeneca Clinical Trials Website AstraZeneca Clinical Trials Website This web site provides clinical trial data, results and other information regarding clinical trials astrazenecagrouptrials.pharmacm.com
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8851R00001&attachmentIdentifier=fae9c38c-734a-468d-84ad-9b52dbfc660f&fileName=D8851R00001-clinical-study-report-synopsis-sanitized.pdf&versionIdentifier=